CLINICAL TRIAL: NCT02525276
Title: Female Sex Hormones, Insulin Resistance and Effects of Exercise in a Human Experimental Model of Menopause
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Rasmussen Rinnov, MD PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-15008066
Record Dates: First submitted 2015-07-29; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- training + HT (Experimental): training + HT
  Interventions: Behavioral: exercise; Drug: Hormone treatment
- training - HT (Experimental): training - HT
  Interventions: Behavioral: exercise
- -training + HT (Placebo Comparator): -training + HT
  Interventions: Drug: Hormone treatment
- - training - HT (No Intervention): - training - HT

INTERVENTIONS:
Behavioral: exercise — The exercise intervention will conduct the following training program 4 days/week for 6 months: endurance training consisting of supervised training on a bike ergometer for 20 min at 70% of maximal heart rate (HR) the first week, increased by 5 min each week until reaching 40 min. Then the intensity will be increased to 80% of max HR over the next month and recalculated every month.
  Arms: training + HT; training - HT
Drug: Hormone treatment — Continually estradiol and gestagens - tablets and patches or cyclic estradiol and gestagens - tablets or patches.
  Including:
  Drospirenon, Norethisteronacetat, Medroxyprogesteronacetat
  Arms: -training + HT; training + HT

SUMMARY:
The main objective of this study is to investigate the role of female sex hormones in relation to insulin resistance in a controlled human experimental model of menopause and to explore whether exercise and/or hormone treatment (HT) can compensate for loss of endogenous sex hormone production by maintaining insulin sensitivity and metabolic activity at a level equivalent to what is seen in premenopausal women.

Loss of ovarian function is associated with an increased incidence of metabolic disease including metabolic syndrome, type 2 diabetes and cardiovascular disease. This increased disease incidence seems to be related to changes in body composition including decreased skeletal muscle mass and increased visceral fat mass as well as decreased whole body fat oxidation and energy expenditure. Regular physical activity decreases general mortality among other things by increasing fat free mass and insulin sensitivity and hereby prevents metabolic syndrome and cardiovascular disease - conditions seen with an increased incidence after menopause and could therefore be a possible treatment.

In the present study the Investigators will assess the role of sex hormones in a model of menopause where healthy women are undergoing planned bilateral oophorectomy due to risk of hereditary ovary cancer. The use of this model makes it possible to control the time point for loss of ovarian function and hereby investigate the timeframe and possible contributing factors in a strictly controlled model. 48 premenopausal women will be included in the study. The study is conducted in women who have already been offered surgical oophorectomy. The first 2 months the study will be an observational cohort study. Hereafter the patients will be allocated to one of four groups (n=12) in a randomized controlled trial, addressing the effects of 6 months of exercise with or without HT. Type of surgery has been decided before inclusion based on medical indications. The women will be offered HT according to national guidelines, but the choice is up to them. Randomization applies only to the training intervention.

Firstly the Investigators aim at investigating the role of endogenous female sex hormones and HT in relation to insulin resistance, whole body fat oxidation and -energy expenditure, changes in visceral fat mass and fat free mass after oophorectomy. Secondly, the Investigators wish to study the molecular mechanisms behind the oophorectomy-induced insulin resistance with a focus on insulin signaling in skeletal muscle and fat tissue. Lastly, the investigators aim to explore whether exercise and/or HT can compensate for loss of endogenous female sex hormone production by maintaining IS and metabolic activity, hereby preventing future incidents of metabolic disease in relation to menopause.

All in all, this project will contribute with new knowledge concerning the question of how endogenous female sex hormones affect insulin sensitivity and metabolic functioning and how exercise may be used as a disease preventive modality for middle-aged women.

ELIGIBILITY:
Inclusion Criteria:

* women
* going through oophorectomy to prevent hereditary cancer
* premenopausal

Exclusion Criteria:

* infection during the last month
* chronic disease
* smoking
* alcohol > 14 servings/week
* hysterectomized
* premature menopause
* BMI > 30

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
insulin sensitivity | 1 year
  Measured by a hyperinsulinemic euglycemic clamp as AUC for glucose infusion rate

CONTACTS AND LOCATIONS:
Overall Officials: Julie Abildgaard, MD, Principal Investigator — Centre of Inflammation and Metabolism